CLINICAL TRIAL: NCT00188552
Title: A Phase II Study of the Use of Pentoxifylline and Vitamin E in the Treatment of Late Radiation Related Injuries
Brief Title: The Use of Pentoxifylline and Vitamin E in the Treatment of Late Radiation Related Injuries
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: May 2007: No annual renewal
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 01-0244-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries | interventions — Pentoxifylline; alpha-Tocopherol

INTERVENTIONS:
Drug: pentoxifylline
Drug: α-Tocopherol

SUMMARY:
Patients with radiation induced injuries experience significant pain and negative effects on quality of life. Currently, no standard therapy for these patients exists, with some patients treated symptomatically, and others treated with hyperbaric oxygen or pentoxifylline/Vitamin E. This study will examine prospectively the safety and efficacy of using a regimen of pentoxifylline and vitamin E in patients with late radiation induced injuries.

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented symptomatic radiation induced injury (e.g. fibrosis, necrosis, ulceration)
* Prior treatment with radiation therapy to the affected area - completed at least 3 months prior to study entry
* Pain in irradiated volume after 3 months (not attributable to acute inflammation)
* ECOG performance status must be 0, 1 or 2
* Life expectancy is greater than 6 months
* Age 18 to 75 years; informed consent

Exclusion Criteria:

* Patient is still responding to other therapies for soft tissue injury
* Active malignant disease
* Any medical illness or condition judged likely by the local investigator to preclude safe administration of protocol treatment, including but not limited to, acute myocardial infarction, severe coronary artery disease, active internal bleeding or a history of hemorrhagic diathesis, peptic ulcer, impaired kidney or liver function
* Pregnant or lactating women
* No contraindication to treatment with pentoxifylline. (i.e. previously exhibited intolerance to pentoxifylline or other xanthines such as caffeine, theophylline or theobromine, recent cerebral and/or retinal hemorrhage)
* Concurrent treatment with warfarin or other anticoagulant, or with erythromycin
* Concurrent treatment with other experimental agents or other treatment for fibrosis
* Patients treated with radiotherapy for breast cancer 3 months to 3 years prior to study entry
* Blood pressure < 90/60 mm Hg or orthostatic hypotension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2002-07

PRIMARY OUTCOMES:
To examine the effect of the combination of Pentoxifylline (Trental™) and α-Tocopherol (Vitamin E) on symptomatic radiation induced fibrosis.

SECONDARY OUTCOMES:
To examine the effect of the combination of Pentoxifylline (Trental™) and α-Tocopherol (Vitamin E) on quality of life in patients with radiation induced fibrosis
To examine the effect of the combination of Pentoxifylline (Trental™) and α-Tocopherol (Vitamin E) on other patient outcomes, including:
ECOG Performance status
To identify factors which modify patients' response to protocol therapy (e.g. radiotherapy treatment factors, prior surgeries, chemotherapy, patient characteristics, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Levin, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada